CLINICAL TRIAL: NCT00872976
Title: Phase 1 Trial of Dasatinib and Bendamustine in Chronic Lymphocytic Leukemia
Brief Title: Study of Dasatinib and Bendamustine in Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Objectives Changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-182
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Dasatinib; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort #1 (Experimental)
  Interventions: Drug: Dasatinib; Drug: Combination of Bendamustine + Dasatinib
- Cohort #2 (Experimental)
  Interventions: Drug: Dasatinib; Drug: Combination of Bendamustine + Dasatinib

INTERVENTIONS:
Drug: Dasatinib — One Week Initial Treatment for Cohort #1: Dasatinib - Tablets/Oral Solution, at assigned dose level, once daily (QD)
  Other Names: BMS-354825; Sprycel
  Arms: Cohort #1
Drug: Combination of Bendamustine + Dasatinib — Dasatinib, Tablets/Oral Solution, Oral, 50 mg, then at 80 mg, at 80 mg, and at 100 mg, once daily (QD), at assigned ascending dose, for 28 day cycles for a maximum of six cycles
  Bendamustine, injection, IV injection, 50 mg/m²/Day 1 and Day 2, then at 50 mg/m², at 70 mg/m², at 70 mg/m², at assigned ascending dose, once daily 30 minute IV infusion Day 1 and Day 2 for a maximum of six cycles
  Other Names: Sprycel; Treanda
  Arms: Cohort #1
Drug: Dasatinib — One Week Initial Treatment for Cohort #2: Dasatinib - Tablets/Oral Solution, at 100 mg, once daily (QD)
  Other Names: BMS-354825; Sprycel
  Arms: Cohort #2
Drug: Combination of Bendamustine + Dasatinib — Dasatinib, Tablets/Oral Solution, Oral, at 100 mg, once daily (QD), for 28 day cycles for maximum of six cycles
  Bendamustine, injection, IV injection, 100 mg/m²/Day 1 and Day 2, once daily 30 minute IV infusion Day 1 and Day 2 for maximum of six cycles
  Other Names: Treanda; Sprycel
  Arms: Cohort #2

SUMMARY:
The purpose of this study is to determine the recommended dose for the combination of dasatinib and bendamustine in chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria (Cohort #1):

* Diagnosis of B-CLL by NCI criteria
* Require chemotherapy and have fully recovered from previous administered chemotherapy
* Subjects must have progressed, failed to achieve a meaningful response, or relapsed/intolerant to prior therapy. Failing at least one purine analogue regimen
* Subjects have received three or fewer prior treatment regimens
* ECOG status of 0 - 2

Inclusion Criteria (Cohort #2):

* If dose level + 3 is reached, the criteria is the same as outlined for Cohort #1, however the subjects should not have a history of prior chemotherapy (treatment naive)

Exclusion Criteria:

* Unwilling or unable to use an acceptable method to avoid pregnancy
* Uncontrolled or significant cardiovascular disease, including prolonged QTc interval
* History of significant bleeding disorder, unrelated to CLL
* Prior concurrent malignancy
* Drugs that generally accepted to have the risk of causing Torsades de Pointes
* Autoimmune hemolytic anemia requiring therapy or transfusion support
* Autoimmune thrombocytopenia requiring steroid therapy or transfusion support
* Richter's Syndrome
* Transformation to prolymphocytic leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) as assessed by measuring dose limiting toxicities (DLT) at each dosing level | From initial dose to the end of three cycles of treatment at each dosing level. Each cycle is 28 days, so approximately 91 days

SECONDARY OUTCOMES:
All response evaluable subjects Cohorts #1 and #2 are assessed for overall response rate(s): complete remission (CR); CR with incomplete marrow recovery (CRi); partial remission (PR); for progressive disease (PD) or stable disease (SD) | From initial dose to the end of six cycles of treatment. Each cycle is 28 days, so approximately 175 days
The effects of treatment on various biological correlates will also be assayed | From initial dose to the end of six cycles of treatment. Each cycle is 28 days, so approximately 175 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution, New Hyde Park, New York
  - Local Institution, Columbus, Ohio
  - Local Institution, Nashville, Tennessee

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx